CLINICAL TRIAL: NCT05383703
Title: A Phase I Clinical Study on Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of MNC-168 Enteric-coated Capsules in Patients With Advanced Malignant Solid Tumors
Brief Title: Clinical Study of MNC-168 Enteric-coated Capsule in the Treatment of Advanced Intestinal Solid Tumor
Acronym: MNC-168
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moon (Guangzhou) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNC-168-101
Record Dates: First submitted 2022-05-05; First posted 2022-05-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-04

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open-label, dose-escalation Phase I clinical trial designed to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of live bacterium MNC-168 as a single oral agent in subjects with advanced malignant solid tumors. To explore the changes of biomarkers and intestinal flora related to curative effect, mechanism of action, safety and/or pathological mechanism.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment of MNC-168 enteric-coated capsules as a single oral drug (Experimental): Treatment of live bacterium MNC-168 as a single oral agent as a single oral drug in subjects with advanced malignant solid tumors. The dosage increased in different stages. Each phase was administered once a day for three weeks.
  Interventions: Drug: Treatment of MNC-168 enteric-coated capsules as a single oral drug

INTERVENTIONS:
Drug: Treatment of MNC-168 enteric-coated capsules as a single oral drug — Treatment of live bacterium MNC-168 as a single oral agent as a single oral drug in subjects with advanced malignant solid tumors. First, live fungi can directly or indirectly inhibit tumor growth or induce tumor cell apoptosis through their metabolites or surface proteins, and can also regulate the immune system, especially the tumor microenvironment, to play an antitumor function. Second, tumor immunotherapies exhibit different response levels in different populations, and live bacterial analogs derived from gut microbes may enhance the response to immunotherapy in weakly responding patients.
  Other Names: Therapy of Live bacteria MNC-168

SUMMARY:
This study is a multicenter, open-label, dose-escalation Phase I clinical trial designed to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of live bacterium MNC-168 as a single oral agent in subjects with advanced malignant solid tumors. To explore the changes of biomarkers and intestinal flora related to curative effect, mechanism of action, safety and/or pathological mechanism.

DETAILED DESCRIPTION:
A total of four dose groups (0.25 × 10^10 colony forming unit, 1 × 10^10 colony forming unit, 5 × 10^10 colony forming unit, and 12.5 × 10^10 colony forming unit) are pre-designed for this study in patients with advanced malignant solid tumors, with three subjects in each dose group in a "3+3" dose escalation design.

ELIGIBILITY:
Subjects must meet all of the following criteria to be included in this study:

1. They voluntarily participate in the clinical study; fully understand, are informed about this study and sign the Informed Consent Form; are willing to follow and have the ability to complete all trial procedures.
2. Subjects are required to meet the following criteria: they must be subjects with histologically or cytologically confirmed advanced malignant solid tumors who do not respond to, or are intolerant to, or reject standard treatment, or receive no effective treatment;
3. ≥18 years old, both male and female;
4. They have an expected survival of ≥ 3 months;
5. Their performance status score is 0 to 1 according to the Eastern Cooperative Oncology Group (ECOG) criteria;
6. There is at least one measurable or assessable lesion according to RECIST V1.1;
7. The organ function must meet the following requirements:

   7.1 No serious hematopoietic abnormalities (no blood transfusion, and no use of blood products, granulocyte colony-stimulating factors, platelet-stimulating factors or other hematopoietic growth factors for correction within 14 days prior to the screening lab test): hemoglobin (HGB) ≥ 90 g/L, neutrophil count (ANC) ≥ 1.5 × 109 /L, platelet count (PLT) ≥ 100 × 109 /L; 7.2 Liver function: alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal (ULN) (subjects without liver metastases) or ≤ 5 × ULN (subjects with liver metastases); serum total bilirubin ≤ 1.5 × ULN, total bilirubin levels in subjects with Gilbert's syndrome ≤ 3.0 × ULN; 7.3 Coagulation function: prothrombin time (PT), international normalized ratio (INR) and partial thromboplastin time (APTT) ≤ 1.5 × ULN; 7.4 Renal function: Creatinine (Cr) ≤ 1.5 × ULN and serum creatinine clearance rate ≥ 50 ml/min (see Appendix 1);
8. Eligible subjects (male or female) of childbearing potential must agree to take a medically approved contraceptive measure (e.g., intrauterine device, pill, or condom) during the trial and for 3 months after the last dose; female subjects of childbearing potential must have a negative pregnancy test result during the screening period and must be non-lactating; See Appendix 2 for specific contraception measures.

Criteria for exclusion

Meeting any 1 of the following exclusion criteria results in exclusion:

1. Subjects are known (including suspected) allergic to the active ingredient MNC-168 or its excipients, or have an allergic constitution (excluding mild asymptomatic seasonal allergies);
2. Subjects have difficulty swallowing or do not tolerate venipuncture or have a history of needle and blood sickness;
3. Toxic reactions from prior antineoplastic therapy have not returned to grade 1 or below (Grade > 1 based on CTCAE 5.0, except for toxicity such as alopecia, which in the judgment of the investigator is not a safety risk);
4. Subjects have bleeding tendencies or are on thrombolytic or anticoagulant therapy.
5. Subjects have received immunosuppressive drugs within 14 days before signing informed consent, except in the following cases:

   5.1 Intranasal, inhalation, topical steroid or topical steroid injection (such as intra-articular injection); 5.2 Systemic corticosteroid therapy with prednisone or its equivalent physiological dose not more than 10 mg/day; 5.3 Use of steroids as prophylactic drugs for allergic reactions (such as pretreatment before computed tomography [CT]).
6. Subjects have received an allogeneic tissue/solid organ transplant;
7. Subjects develop spinal cord compression, brain metastases or meningeal metastases, excluding those who do not need steroid therapy after surgery, whole brain radiotherapy or stereotactic radiosurgery, and whose disease is stable for ≥ 8 weeks and/or ≥ 4 weeks before the first administration;
8. Subjects have had a cerebrovascular accident or a history of transient ischemic attack within 6 months prior to signing the informed consent form;
9. Subjects require systemic antibacterial, antiviral or antifungal therapy for any uncontrolled active infection at the time of signing the informed consent and/or within 1 week prior to Cycle 1 Day 1 (C1D1); and subjects have received a course of systemic antibiotics within 2 weeks prior to C1D1;
10. Subjects have a history of other primary malignancies within 5 years prior to the investigational therapy, with the following exceptions: radically treated malignancies that have not recurred, such as cervical carcinoma in situ, basal cell carcinoma of the skin or squamous cell carcinoma;
11. Subjects have active gastrointestinal diseases or other diseases that may significantly affect the absorption, distribution, metabolism or excretion of MNC-168;
12. Subjects have a clear history of neurological or psychiatric disorders (including epilepsy and dementia);
13. Subjects have received chemotherapy, radiotherapy or biological anticancer therapy, herbal therapy with antitumor effects, and palliative local radiotherapy within 2 weeks prior to the first dose;
14. Subjects have taken live biotherapeutic products (LBPs), prebiotic foods and/or beverages and/or supplements (e.g., yogurt) within 1 week prior to the first dose or require regular doses of LBPs, prebiotic foods or supplements during the study period;
15. Subjects have received fecal transplantation, preparation of spores or other fecal materials, isolated bacterial products, genetically engineered bacteria, or similar drug treatment;
16. Subjects have participated in a clinical trial of another investigational drug or investigational device within 4 weeks (or 5 half-lives of the drug, whichever is more appropriate in the judgment of the investigator) prior to the first dose; note: subjects who have entered the follow-up phase of a clinical study may be eligible as long as it has been more than 4 weeks (or 5 half-lives of the drug, whichever is more appropriate in the judgment of the investigator) since the last dose in the previous study;
17. Subjects have undergone major surgical procedures or active ulcers or wounds that have not fully healed within 4 weeks prior to the first dose of the trial; or require major surgical procedures during the trial;
18. Subjects develop peripheral neuropathy ≥ grade 2;
19. Subjects have clinically significant cardiovascular diseases, including any of the following cases:

    19.1 Subjects have a history of myocardial infarction (within 6 months prior to trial), severe or unstable angina, coronary or peripheral artery bypass grafting; 19.2 New York Heart Association (NYHA) grade 3~4 heart failure; 19.3 Cardiac function: left ventricular ejection fraction (LVEF) < 50%. 19.4 Poorly controlled hypertension (systolic blood pressure ≥ 150 mm Hg and/or diastolic blood pressure ≥ 95 mm Hg); 19.5 Subjects are considered by the investigator to have clinically significant arrhythmias or electrocardiographic (ECG) abnormalities, such as the mean of three heart rate-corrected QT intervals (QTcF) intervals of > 470 msec calculated for three 12-lead ECG measurements performed at the investigation site; 19.6 Subjects are currently receiving certain medications that have a known risk of prolonging the QT interval or inducing tip-twist ventricular tachycardia and are unable to discontinue the medication or switch to another medication 1 week prior to the start of treatment with the investigational drug.
20. Subjects were HIV-infected or active hepatitis B virus-infected (HBsAg and/or HBcAb positive with a peripheral blood hepatitis B virus DNA titer test ≥ 1 × 103 IU/ml), or active hepatitis C virus-infected (hepatitis C virus antibody positive with hepatitis C virus RNA ≥ 500 IU/ml);
21. Subjects have received an attenuated/inactivated vaccine within 28 days prior to signing informed consent or are scheduled to receive an attenuated/inactivated vaccine during the screening period;
22. Subjects, in the judgment of the investigator, have a serious concomitant disease that endangers the safety of the subject, or interferes with the subject's ability to complete the study;
23. Subjects are those with a history of psychotropic substance abuse or drug use;
24. Or an investigator has determined that the subject has other conditions that make him/her eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability indexes | 2 years
  The safety is evaluated by The National Cancer Institute Common Terminology Criteria for Adverse Events（NCI-CTCAE）V5.0.

SECONDARY OUTCOMES:
pharmacokinetic index | 2 years
  Total colony forming unit(CFU) of Enterococcus lactis excreted in stools, expressed as raw values and log10 conversion
pharmacokinetic indexes | 2 years
  CFU/g of Enterococcus lactis excreted in stools, expressed as raw values and log10 conversion
Efficacy evaluation indexes | 2 years
  Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 are adopted for solid tumor efficacy evaluation in this study. The guidelines describe a standard method for measuring solid tumors and defining objective changes in tumor size in adult and pediatric tumor clinical trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China